CLINICAL TRIAL: NCT06248294
Title: PRogression Of bicuSPid-rElated aoRtOpathy in Patients Undergoing Transcatheter Aortic Valve Implantation: The PROSPERO-TAVI Multi Center, International Registry
Brief Title: PRogression Of bicuSPid-rElated aoRtOpathy in Patients Undergoing Transcatheter Aortic Valve Implantation (PROSPERO-TAVI)
Acronym: PROSPERO-TAVI
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Catania (Other)
Responsible Party: Principal Investigator, Giuliano Costa, Principal Investigator, University of Catania
Other Study IDs: UCatania003
Record Dates: First submitted 2024-01-20; First posted 2024-02-08 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-01

CONDITIONS: Bicuspid-related Aortopathy; Aortic Stenosis
Keywords: BAV; TAVI; Aortopathy
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TAVI patients with native BAV: Patients undergoing TAVI for severe aortic stenosis and native bicuspid aortic valve
  Interventions: Diagnostic Test: CT follow-up

INTERVENTIONS:
Diagnostic Test: CT follow-up — Computed tomography angiography assessment of BAV-related aorthopathy

SUMMARY:
Transcatheter aortic valve implantation (TAVI) is being offered to younger patients affected by severe aortic stenosis as an alternative to surgery. Although historically excluded from the main randomized clinical trials, patients with native bicuspid aortic valve (BAV) are commonly treated in daily TAVI practice. Indeed, several observational studies reported similar outcomes of TAVI in BAV patients compared to tricuspid aortic valve (TAV) patients. Notably, BAV is frequently associated with aortic dilatation (20% to 84% of BAV patients). Surgical patients usually undergo concomitant aortic root replacement if aortic diameter exceed 50 mm (5). TAVI patients do not undergo treatment of the concomitant aortopathy, but currently there is a paucity of data regarding the progression of the aortopathy after AS treatment (6,7).

The main aim of this ambispective, multicenter study is to evaluate the progression of the bicuspid valve-associated aortopathy in patients undergoing TAVI by computed tomography angiography (CTA) assessment at follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing TAVI with native BAV from January 2018 to December 2019

Exclusion Criteria:

* Patients undergoing TAVI without native BAV
* Patients receiving first generation TAVI device
* Patients undergoing TAVI before January 2018 or after December 2019

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing TAVI for severe aortic stenosis and native bicuspid aortic valve
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Absolute difference in maximum aortic diameters at multiple levels of ascending aorta | 5 years
  Measurements of maximum aortic diameters at follow-up CTA assessment will be compared with values at pre-TAVI CTA assessment

SECONDARY OUTCOMES:
Death, stroke or rehospitalization for heart failure | 5 years
  Death, stroke or rehospitalization for heart failure
Aortic events leading to urgent intervention or elective aortic root replacement | 5 years
  Aortic events (i.e. fissuration, dissection) after the index intervention leading to aortic intervention, or elective aortic root replacement.
Bioprosthesis dysfunction (HALT or RLM at 4-D CTA assessment) | 5 years
  Presence of hypo-attenuated leaflet thickening (HALT)/reduced leaflet motion (RLM) at follow-up four-dimensional CTA assessment

CONTACTS AND LOCATIONS:
Locations (1):
- AOU Policlinico G. Rodolico - San Marco, Catania, Italy

IPD SHARING:
Plan to Share IPD: Undecided